CLINICAL TRIAL: NCT00517244
Title: Child Anxiety Disorders: Parenting and Temperament Effects
Brief Title: Evaluating Parenting Styles and Child Temperament Associated With Child Anxiety Disorders
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Abbe Garcia, Assistant Professor (Research)/Assistant Director Child Outpatient Psychiatry, Rhode Island Hospital
Other Study IDs: K23MH071754 (NIH); K23MH071754 (NIH); DDTR B3-PDX
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Anxiety Disorders; Obsessive Compulsive Disorder
Keywords: Children; Healthy Controls; Assessment
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Primary anxiety disorder
- B: Primary obsessive compulsive disorder
- C: Healthy children with no previous history of an anxiety disorder

SUMMARY:
This study will look at similarities and differences in family processes and child temperament among children with and without symptoms of anxiety disorders.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common childhood disorders. Although anxiety is a normal part of life and growing up, for some children this anxiety becomes chronic, relentless, and progressively worse if left untreated. Physical symptoms typically accompany the intense anxiety caused by the disorder, and may include blushing, profuse sweating, trembling, nausea, and difficulty talking. Effective treatments for anxiety disorders are available, and research continues to yield new, improved therapies that can help most people with anxiety disorders to lead productive, fulfilling lives. This study will look at similarities and differences in family processes and child temperament among children with and without symptoms of anxiety disorders. Results from this study may improve future treatment of children with anxiety disorders.

Families participating in this observational study will be mailed parent and child questionnaires that should be completed prior to the first study session. The child questionnaires will ask for information regarding the child's feelings and family interactions. Parent questionnaires will ask for information about their own personal feelings as well as the child's feelings, symptoms, and behaviors. Study participation will last 2 days. On the first day of the study, families will undergo a 3-hour diagnostic interview in which questions similar to those found on the questionnaires will be revisited. On the second day, mothers and their children will participate in three different observation tasks that explore how families interact and respond to certain situations. These tasks may include discussing certain anxiety-provoking situations, putting puzzles together, and creating an ending to a story. Before each task, the child will be placed alone in a separate room where the child will be asked to relax. Throughout the tasks, the child's heart rate and breathing will be recorded by a machine. The tasks will be videotaped but will be viewed only by research staff for data analysis purposes and to ensure that all safety procedures were followed. Upon study completion, if it appears that a child has an anxiety disorder, parents of the child will be notified and will receive treatment referrals as needed.

ELIGIBILITY:
Inclusion Criteria for Children:

* English-speaking

Exclusion Criteria Children:

* Mental retardation
* Current or past diagnosis of autistic spectrum disorders
* Current or past diagnosis of psychotic disorders

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2006-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Parenting styles and child temperaments associated with child anxiety disorders | Measured at completion of treatment analysis

CONTACTS AND LOCATIONS:
Overall Officials: Abbe M. Garcia, PhD, Principal Investigator — Brown Medical School/ Rhode Island Hospital
Locations (1):
- Pediatric Anxiety Research Center/Bradley Hospital/Brown Medical School, Providence, Rhode Island, United States